CLINICAL TRIAL: NCT03267173
Title: Evaluate the Safety and Efficacy of Chimeric Antigen Receptor Engineered T Cell Immunotherapy (CAR-T) in the Treatment of Pancreatic Cancer in a Single Center, Non Controlled Clinical Study.
Brief Title: Evaluate the Safety and Efficacy of CAR-T in the Treatment of Pancreatic Cancer.
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Harbin Medical University (Other)
Collaborators: Shanghai Unicar-Therapy Bio-medicine Technology Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Yunwei Wei
Record Dates: First submitted 2017-08-27; First posted 2017-08-30 (Actual); Last update posted 2017-08-30 (Actual); Status verified 2017-08

CONDITIONS: Pancreatic Cancer; CAR
Keywords: Pancreatic Cancer; CAR-T; Mesothelin; CEA; HER2
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAR-T (Experimental): A single dose of Chimeric antigen receptor T cells will be administered by vascular interventional mediated as one dose infusions. According to the patient's condition and weight, the intervention dose of aE7 CAR-T cells per kilogram of body weight was treated once.
  Interventions: Drug: Chimeric antigen receptor T cell

INTERVENTIONS:
Drug: Chimeric antigen receptor T cell — Evaluate the efficacy and safety of targeted Mesothelin/PSCA/CEA/HER2/MUC1/, EGFRvIII and other chimeric antigen receptor engineered T cell immunotherapy in the treatment of pancreatic cancer.
  Other Names: meso-CAR

SUMMARY:
Immunotherapy has become the major breakthrough and the most promising treatment, with the host of development of tumor biology, molecular biology and immunology. It has become the fourth tumor treatment model after traditional tumor therapies (surgery, chemotherapy, radiotherapy) . Mesothelin, PSCA, CEA, HER2, MUC1 and EGFRvIII are potential targets and spectacular paradigm in the diagnosis and treatment of pancreatic cancer. This study is for evaluation of the safety and efficacy of Mesothelin, PSCA, CEA, HER2, MUC1, EGFRvIII targeted and other CAR-T cell immunotherapy for pancreatic cancer.

DETAILED DESCRIPTION:
Immunotherapy has become the major breakthrough and the most promising treatment, with the host of development of tumor biology, molecular biology and immunology. It has become the fourth tumor treatment model after traditional tumor therapies (surgery, chemotherapy, radiotherapy) . With the development of the research field, the CAR-T cell basis and clinical research of various targets have achieved good results. Mesothelin, PSCA, CEA, HER2, MUC1 and EGFRvIII are potential targets and spectacular paradigm in the diagnosis and treatment of pancreatic cancer. This study is for evaluation of the safety and efficacy of Mesothelin, PSCA, CEA, HER2, MUC1, EGFRvIII targeted and other CAR-T cell immunotherapy for pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Imaging, pathology or biopsy confirmed as pancreatic cancer and it has metastasized, can not radical cured by surgery; patients restored good but there is still residual lesions, recurrence or metastasis 1 months after surgery;
* Accepted more than 1 times chemotherapy which is invalid or unwilling to accept previous chemotherapy patients;
* The corresponding antigens such as Meso and PSCA/ CEA/ HER2/ MUC1/ EGFRvIII were highly expressed;
* Male patients aged between 18 and 65;
* Life expectancy greater than 1 months;
* Karnofsky score ≥ 60, ECOG≤ 2;
* Important organ function as defined by the following: cardiac ejection fraction ≥ 50%; electrocardiogram showed no obvious abnormalities; creatinine clearance rate calculated by using Cockcroft- Gault formula ≥40ml/min ; ALT/AST≤ 3×the institution normal upper limit; total bilirubin ≤2.0mg/dl; coagulation function: PT/ APPT<2 ×the institution normal upper limit; SpO2 >92%; Blood: hemoglobin>80g/L, ANC ≥ 1, PLT ≥ 50×109/L;
* There is measurable target lesion;
* Voluntary informed consent is given.

Exclusion Criteria:

* Immunosuppressive drugs or hormones were used a week before admission;
* Severe active infection;
* Human immunodeficiency virus (HIV) positive;
* Active hepatitis B or C infection;
* Past medical history of other malignancies. Not included: patients who have been cured at any time prior to the treatment of the skin basal or squamous cell carcinoma and cervical carcinoma in situ; the other tumor has not listed above, but has been used and only cured by surgery, without further treatment by other measures, the subjects of disease-free survival more than 5 years, can be included in the study;
* Patients participating in other clinical trials;
* The researchers thought the subjects were unfit for inclusion or unable to participate in or complete the study；
* Patients with congenital immunodeficiency；
* There is a history of myocardial infarction and serious arrhythmia within six months.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2017-06-15 (Actual); Primary Completion 2019-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Number of patients with tumor response | 8 weeks
  Tumor response is assessmented with Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1

SECONDARY OUTCOMES:
Number of patients with adverse event | 8 weeks
  Asverse event is evaluated with CTCAE, version 4.0

CONTACTS AND LOCATIONS:
Overall Officials: Wei Yunwei, Dctor, Study Director — First Affiliated Hospital of Harbin Medical University
Locations (1):
- Harbin Medical University, Harbin, Heilongjiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zervos E, Agle S, Freistaedter AG, Jones GJ, Roper RL. Murine mesothelin: characterization, expression, and inhibition of tumor growth in a murine model of pancreatic cancer. J Exp Clin Cancer Res. 2016 Mar 1;35:39. doi: 10.1186/s13046-016-0314-2. PMID 26931187
- [Background] Freedman JD, Hagel J, Scott EM, Psallidas I, Gupta A, Spiers L, Miller P, Kanellakis N, Ashfield R, Fisher KD, Duffy MR, Seymour LW. Oncolytic adenovirus expressing bispecific antibody targets T-cell cytotoxicity in cancer biopsies. EMBO Mol Med. 2017 Aug;9(8):1067-1087. doi: 10.15252/emmm.201707567. PMID 28634161
- [Background] Morello A, Sadelain M, Adusumilli PS. Mesothelin-Targeted CARs: Driving T Cells to Solid Tumors. Cancer Discov. 2016 Feb;6(2):133-46. doi: 10.1158/2159-8290.CD-15-0583. Epub 2015 Oct 26. PMID 26503962
- [Background] Le DT, Wang-Gillam A, Picozzi V, Greten TF, Crocenzi T, Springett G, Morse M, Zeh H, Cohen D, Fine RL, Onners B, Uram JN, Laheru DA, Lutz ER, Solt S, Murphy AL, Skoble J, Lemmens E, Grous J, Dubensky T Jr, Brockstedt DG, Jaffee EM. Safety and survival with GVAX pancreas prime and Listeria Monocytogenes-expressing mesothelin (CRS-207) boost vaccines for metastatic pancreatic cancer. J Clin Oncol. 2015 Apr 20;33(12):1325-33. doi: 10.1200/JCO.2014.57.4244. Epub 2015 Jan 12. PMID 25584002
- [Background] Abate-Daga D, Lagisetty KH, Tran E, Zheng Z, Gattinoni L, Yu Z, Burns WR, Miermont AM, Teper Y, Rudloff U, Restifo NP, Feldman SA, Rosenberg SA, Morgan RA. A novel chimeric antigen receptor against prostate stem cell antigen mediates tumor destruction in a humanized mouse model of pancreatic cancer. Hum Gene Ther. 2014 Dec;25(12):1003-12. doi: 10.1089/hum.2013.209. PMID 24694017
- See also: References are all derived from PubMed — http://www.ncbi.nlm.nih.gov